CLINICAL TRIAL: NCT04753125
Title: Interventions for Enhancing Adherence to Syphilis Treatment and Follow-up: Study Protocol for the Health Information and Monitoring of Sexually Transmitted Infections (SIM) Randomized Controlled Trial
Acronym: SIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Vanessa Martins de Oliveira, Prof Eliana Marcia Ross Wendland, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000001
Record Dates: First submitted 2021-01-28; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Syphilis
Keywords: Prevalence; Incidence; Men who have sex with men; Protocol
MeSH Terms: conditions — Syphilis; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- compliance treatment (Active Comparator): controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance for 3, 6. 9 and 12 months
  Interventions: Behavioral: follow-up by telephone; Behavioral: follow-up via a game in a smartphone app; Behavioral: conventional follow-up by a health professional
- compliance for blood test (Active Comparator): controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance, follow-up via a game in a smartphone app through an interactive game with stimuli to pass the phase as the treatment was completed and blood tests were performed in 3,6,9 and 12 months.
  Interventions: Behavioral: follow-up by telephone; Behavioral: follow-up via a game in a smartphone app; Behavioral: conventional follow-up by a health professional
- demographic socio-economic and sexuality questionnaire (Placebo Comparator): Questionnaire applied to all patients with positive VDRL
  Interventions: Behavioral: follow-up by telephone; Behavioral: follow-up via a game in a smartphone app; Behavioral: conventional follow-up by a health professional

INTERVENTIONS:
Behavioral: follow-up by telephone — The SIM study is a single-centre, randomized, controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance
Behavioral: follow-up via a game in a smartphone app — The SIM study is a single-centre, randomized, controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance
Behavioral: conventional follow-up by a health professional — The SIM study is a single-centre, randomized, controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance

SUMMARY:
The SIM study is a single-centre, randomized, controlled trial with a 12-month follow-up period. The aim is to determine which of the 3 methods of follow-up is the most effective in promoting patient treatment compliance. The recruitment of participants will be done by invitation, and tests will be performed in a mobile unit in locations accessible to large populations. The goal is to perform 10,000 quick tests, with results confirmed by venereal disease research laboratory (VDRL) tests. Patients with a confirmed diagnosis according to VDRL test results will be randomized in one of three monitoring arms: follow-up by telephone, follow-up via a game in a smartphone app, or conventional follow-up by a health professional. All analyses will follow the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* All adults aged 18 years and older with sorologic test positive for syphilis

Exclusion Criteria:

* Participants who did not return after three contact attempts will be excluded from the study,
* pregnant women
* participants who are not able to provide contact information
* participants who are illiterate
* participants those who underwent syphilis treatment within the previous three months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All adults aged 18 years and older
Enrollment: 10000 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
complince of treatment | ut to 12 months (July 2023)
  3 doses of penicillin g benzathine 3,000,000 UI. The injections are given in the gluteal region once a week from the first dose.
complince of exams | up to 12 months (July 2023)
  Performing the VDRL blood test that should be done at 3, 6, 9 and 12 months after treatment with penicillin.

SECONDARY OUTCOMES:
identify behavioral risk factors for non-adherence to treatment | upt to 12 months (July 2023)
  Identification of risk factors for non-adherence to treatment that will be carried out using a questionnaire applied to study participants with social, racial, sexual, economic and demographic issues.

IPD SHARING:
Plan to Share IPD: Undecided